CLINICAL TRIAL: NCT00784862
Title: A Randomised, Double Blind Trial to Assess the Pharmacokinetics of Arimidex Alone, Nolvadex Alone, or Arimidex and Nolvadex in Combination, When Used as Adjuvant Treatment for Breast Cancer in Postmenopausal Women
Brief Title: ATAC - Pharmacokinetics (PK) Sub-Protocol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Francisco Sapunar, Medical Science Director, Arimidex and Faslodex, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1033IA/0029; D5392C02301
Record Dates: First submitted 2008-11-03; First posted 2008-11-04 (Estimated); Last update posted 2009-05-15 (Estimated); Status verified 2009-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Arimidex 1mg + Nolvadex placebo
  Interventions: Drug: Anastrozole
- 2 (Active Comparator): Arimidex placebo + Nolvadex 20mg
  Interventions: Drug: Anastrozole; Drug: Tamoxifen
- 3 (Active Comparator): Arimidex 1mg + Nolvadex 20mg
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Anastrozole — 1mg, orally, once daily
  Other Names: Arimidex
  Arms: 1; 2
Drug: Tamoxifen — 20mg, orally, once daily
  Other Names: Nolvadex
  Arms: 2; 3

SUMMARY:
To assess the effect of ARIMIDEX on the pharmacokinetics of tamoxifen and the effects of tamoxifen on the pharmacokinetics of ARIMIDEX..

ELIGIBILITY:
Inclusion Criteria:

* Eligible for entry into the main ATAC trial 1033IL/0029
* Patients must have been taking ATAC trial medication for at least 3 months (i.e. patients must have reached at least visit 2 of the main ATAC study)
* Patients should be taking their medication in the mornings for at least 3 months
* Patients must be 100% compliant over the preceding fourteen days

Exclusion Criteria:

* Excluded from entry into the main ATAC trial (1033IL/0029)
* Patients whose concurrent treatment includes diazepam or drugs which might affect tamoxifen steady state levels or steroid hormone status. These include ketoconazole (antifungal) or related compounds

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9358 (Actual)
Dates: Start 1998-06; Study Completion 1999-03 (Actual)

PRIMARY OUTCOMES:
Steady state plasma trough concentrations of tamoxifen, desmethyltamoxifen and anastrozole | 24±4 hours after previous dose